CLINICAL TRIAL: NCT07067164
Title: Clinical Performance of Highly Viscous Glass Ionomer Versus Bulk Fill Resin Composite Restorative Materials in Moderate Class II Cavities of Permanent Posterior Teeth " A 12-Month Randomized Clinical Study"
Brief Title: Clinical Performance of HVGIC vs Bulk Fill Composite in Class II Cavities of Posterior Teeth: A 12-Month RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OPD 24 32 (D); 122301 (Other: FDASU-REC)
Record Dates: First submitted 2025-07-05; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-02

CONDITIONS: Comparison of Bulk Fill vs HVGIC in Class II Cavities
Keywords: Bulk fill resin composite; Highly viscous glass ionomer; Class II cavities; Randomized clinical trial; Split-mouth design

STUDY DESIGN:
Intervention Model Description: This study utilizes a split-mouth crossover design in which each participant receives both interventions-bulk fill resin composite and highly viscous glass ionomer restorations-randomly assigned to contralateral moderate Class II cavities. This intra-individual comparison minimizes confounding variables and allows direct evaluation of the clinical performance of each material under similar oral conditions.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were unaware of which material was used on each side of the mouth (participant blinding). Two independent, calibrated outcome assessors who were not involved in the treatment procedures and blinded to the allocation evaluated the restorations using the modified USPHS criteria at each follow-up interval.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bulk Fill Resin Composite (Experimental): Moderate Class II cavities in permanent posterior teeth restored using bulk fill resin composite material, following selective enamel etching and adhesive application under rubber dam isolation, according to the manufacturer's instructions.
  Interventions: Other: Bulk fill resin composite restorative material
- Highly Viscous Glass Ionomer (Experimental): Contralateral moderate Class II cavities in permanent posterior teeth restored using highly viscous glass ionomer material, after cavity conditioning with polyacrylic acid under cotton roll isolation, following manufacturer's instructions
  Interventions: Other: Bulk fill resin composite restorative material

INTERVENTIONS:
Other: Bulk fill resin composite restorative material — Both restorative materials were applied in a clinical setting following standard infection control protocols and material-specific preparation techniques. The interventions were performed by the same calibrated operator to ensure consistency, and evaluated using modified USPHS criteria by two blinded, independent assessors at 1 week (baseline), 6 months, and 12 months. The study employed a split-mouth design to allow direct intra-individual comparison between the two materials under similar oral conditions.
  Other Names: Highly viscous glass ionomer restorative material

SUMMARY:
Study Title:

Clinical Performance of Highly Viscous Glass Ionomer versus Bulk Fill Resin Composite Restorative Materials in Moderate Class II Cavities of Permanent Posterior Teeth: A 12-Month Randomized Clinical Study

Study Design:

Split-mouth, randomized clinical trial on 31 patients with at least two moderate Class II carious lesions in permanent posterior teeth. Each patient receives two restorations-bulk fill resin composite on one side and highly viscous glass ionomer (HVGIC) on the other.

Aim:

To compare the clinical performance of bulk fill resin composite and HVGIC restorations over 1 week (baseline), 6 months, and 12 months using the modified United States Public Health Services (USPHS) criteria.

Primary Outcome:

Marginal adaptation of the restorations

Secondary Outcomes:

1. Anatomic form
2. Contact point
3. Restoration retention
4. Marginal discoloration
5. Surface texture
6. Color match
7. Secondary caries
8. Postoperative sensitivity

Methodology Highlights:

Evaluation by two blinded examiners

Standardized cavity prep and material application

Clinical evaluation using USPHS criteria at all follow-up intervals

Statistical analysis with chi-square, ANOVA, or non-parametric tests as appropriate (R software v4.3.2)

Ethical Considerations:

Approved by the Faculty of Dentistry, Ain Shams University Research Ethics Committee

Informed consent will be obtained from all participants

Significance:

This study helps determine whether HVGIC can be a clinically viable alternative to bulk fill resin composite in moderate Class II cavities, with implications for durability, patient compliance, and cost-effectiveness

DETAILED DESCRIPTION:
Title:

Clinical Performance of Highly Viscous Glass Ionomer versus Bulk Fill Resin Composite Restorative Materials in Moderate Class II Cavities of Permanent Posterior Teeth: A 12-Month Randomized Clinical Study

Study Overview:

This study is a prospective, randomized, split-mouth clinical trial designed to compare the clinical performance of bulk fill resin composite and highly viscous glass ionomer (HVGIC) restorative materials in moderate Class II cavities of permanent posterior teeth over a 12-month period. The evaluation of restorations will be based on the modified United States Public Health Services (USPHS) criteria at three time intervals: 1 week (baseline), 6 months, and 12 months post-treatment.

Rationale and Background:

The challenge of achieving a long-lasting, mechanically resilient, esthetically acceptable restoration in stress-bearing areas such as Class II cavities continues to drive innovation in restorative dentistry. While resin composites offer favorable physical and esthetic properties, their inherent polymerization shrinkage and technique sensitivity have prompted the development of alternatives like bulk fill composites, which allow deeper curing and reduced shrinkage. Meanwhile, glass ionomer materials-notably HVGICs-have seen advancements aimed at improving their physical and mechanical properties, particularly with the introduction of resin coating systems such as the EQUIA system. The need for comparative clinical evaluation under real-world conditions remains critical to guide clinical decision-making.

Aim of the Study:

To evaluate and compare the clinical performance of bulk fill resin composite and highly viscous glass ionomer restorations in moderate Class II cavities of permanent posterior teeth over time using the modified USPHS evaluation criteria.

Objectives:

To assess the clinical behavior of bulk fill resin composite and HVGIC restorations in Class II cavities.

To determine the effect of time (1 week, 6 months, and 12 months) on the clinical performance of these restorative materials.

Research Question:

Is there a significant difference in the clinical performance between bulk fill resin composite and highly viscous glass ionomer restorations in moderate Class II cavities of permanent teeth over a 12-month follow-up?

Hypothesis:

The null hypothesis (H₀) states that there is no significant difference in clinical performance between the two restorative materials, nor does the time interval significantly influence their performance.

Study Design:

A split-mouth, randomized controlled clinical trial involving 31 patients, each presenting with at least two moderate Class II carious lesions, one on each side of the mouth. This design allows direct intra-individual comparison between materials under similar oral conditions.

Setting:

Outpatient clinics of the Operative Dentistry Department, Faculty of Dentistry, Ain Shams University, Cairo, Egypt.

Sample Size Calculation:

Based on a power analysis with α = 0.05, β = 0.2 (power = 80%), and an effect size of ω = 0.398, the calculated sample size was 62 restorations (31 patients). A 15% increase was added to account for possible dropouts, resulting in a final sample of 72 restorations (36 patients).

Randomization and Blinding:

Random allocation will be performed using www.randomization.com. Allocation concealment will be ensured, and two independent blinded evaluators will perform outcome assessment at each follow-up point.

Clinical Procedure:

Bulk fill composite group: Rubber dam isolation, selective enamel etching, universal adhesive application, placement of bulk fill composite per manufacturer's instructions.

HVGIC group: Cotton roll isolation, cavity conditioning with polyacrylic acid, insertion of HVGIC using a capsule system, finishing with diamond stones on the same day.

Follow-up and Evaluation:

Clinical evaluation at 1 week, 6 months, and 12 months using the modified USPHS criteria, which include:

Statistical Analysis:

Categorical data: Chi-square test

Numerical and ordinal data: Shapiro-Wilk test for normality

If normally distributed: Repeated measures ANOVA with Bonferroni post hoc test

If not: Friedman's test with Dunn's post hoc

Significance level: p < 0.05

Software: R version 4.3.2 for Windows

Ethical Considerations:

Study approved by the Faculty of Dentistry, Ain Shams University Research Ethics Committee

Participants will provide informed written consent

No harm expected beyond standard dental procedures; restorations needing repair or replacement will be redone free of charge

Funding:

No external funding was received.

Risks and Benefits:

Risks:

Minimal: possible restoration failure requiring repair or replacement

Benefits:

Free treatment and 12-month follow-up

Improved understanding of restorative options for clinicians and patients

Research Significance:

This study provides valuable clinical data comparing two widely used restorative materials under routine conditions. The findings may influence material selection in moderate Class II cavities and support evidence-based improvements in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 45 years
2. Systemically healthy individuals
3. Patients with at least two Class II carious lesions (one on each side) in permanent posterior teeth
4. Vital, symptomless teeth
5. Teeth in occlusion and in contact with adjacent natural teeth
6. Healthy periodontal tissues
7. Carious lesions of moderate depth (outer or middle third of dentin radiographically)
8. Patients likely to return for recall visits

Exclusion Criteria:

1. Medically compromised patients
2. Pregnant or breastfeeding women
3. Poor oral hygiene
4. Patients undergoing orthodontic treatment
5. Patients with parafunctional habits (e.g., bruxism)
6. Extensive lesions requiring cusp coverage
7. Absence of adjacent or opposing teeth

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Marginal adaptation of the restoration | 1 week (baseline), 6 months, and 12 months after restoration
  Clinical evaluation of the marginal adaptation of bulk fill resin composite and highly viscous glass ionomer restorations in moderate Class II cavities using the modified United States Public Health Service (USPHS) criteria. Marginal adaptation will be scored as Alfa (no gap), Bravo (visible defect without dentin exposure), or Charlie (failure with dentin exposure)

SECONDARY OUTCOMES:
Anatomic form of the restoration | 1 week (baseline), 6 months, and 12 months after restoration
  Clinical evaluation of the anatomical form of restorations using modified USPHS criteria (Alfa: continuous, Bravo: small discontinuity, Charlie: loss of material
Contact point integrity | 1 week (baseline), 6 months, and 12 months after restoration
  Assessment of interproximal contact point using USPHS criteria (Alfa: normal or no contact without irritation, Charlie: no contact with periodontal irritation).
Restoration retention | 1 week (baseline), 6 months, and 12 months after restoration
  Evaluation of whether restorations are fully retained or partially/completely lost using USPHS retention criteria
Marginal discoloration | 1 week (baseline), 6 months, and 12 months after restoration
  Evaluation of marginal staining or discoloration using USPHS scores (Alfa, Bravo, Charlie).
Surface texture | 1 week (baseline), 6 months, and 12 months after restoration
  Clinical assessment of restoration surface texture using an explorer and USPHS criteria (smooth, rough, porous)
Color match | 1 week (baseline), 6 months, and 12 months after restoration
  Evaluation of restoration color and translucency in comparison to adjacent tooth structure using USPHS criteria.
Presence of secondary caries | 1 week (baseline), 6 months, and 12 months after restoration
  Visual and tactile examination to detect recurrent caries adjacent to the restoration using USPHS criteria.
Postoperative sensitivity | 1 week (baseline), 6 months, and 12 months after restoration
  Patient-reported sensitivity following restoration placement, assessed as present or absent.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Kamel, PhD, Principal Investigator — Associate Professor of Operative Dentistry Faculty of Dentistry Ain Shams University
Locations (1):
- Faculty of Dentistry, Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No